CLINICAL TRIAL: NCT03723265
Title: Personalized CRT - Product Surveillance Registry (PSR)
Brief Title: Personalized CRT - PSR
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Personalized CRT
Record Dates: First submitted 2018-10-15; First posted 2018-10-29 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy

SUMMARY:
The purpose of this study is to evaluate the cardiac resynchronization therapy (CRT) response in a real-world patient population and evaluate options to address non-response and patient management.

DETAILED DESCRIPTION:
The Personalized CRT study is a multi-center, single arm, prospective observational study. The purpose of the study is to better understand and characterize heart failure (HF) patient management by characterizing the use and clinical benefit of Medtronic market-released features/tools within the HF Patient Management portfolio.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive or be treated with an eligible CRT device
* Patient within 30 days of therapy received at the time of their initial PSR platform enrollment

Exclusion Criteria:

* Patient who is, or is expected to be inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/ or device study that may confound results

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients that are or will be implanted with an eligible CRT system.
Sampling Method: Non-Probability Sample
Enrollment: 1517 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
CRT Response | Every 3-9 months
  A Clinical Composite Score (CCS) endpoint will be used to assess a change in CRT response for all patients from baseline to follow-up visits.

SECONDARY OUTCOMES:
Treatments for CRT non-response | Every 3-9 months
  Summary statistics will be obtained to describe the distribution of different treatments (or no treatment) the patient receives.
Treatment effects for different CRT features in the CRT non-responder population | Every 3-9 months
  A Clinical Composite Score (CCS) endpoint will be used to assess a change in CRT response.
Patient outcome post initial CRT implant | Every 3-9 months
  Patient outcome will be measured as the patient first occurrence of HF related hospitalization or death.

CONTACTS AND LOCATIONS:
Locations (122):
- United States (88):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Gilbert, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - Palm Springs, California
  - Rancho Mirage, California
  - Redwood City, California
  - Salinas, California
  - San Diego, California
  - Stanford, California
  - Torrance, California
  - Van Nuys, California
  - Denver, Colorado
  - Lakewood, Colorado
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Clearwater, Florida
  - Jacksonville, Florida
  - Safety Harbor, Florida
  - Albany, Georgia
  - Marietta, Georgia
  - Evansville, Indiana
  - Indianapolis, Indiana
  - West Des Moines, Iowa
  - Kansas City, Kansas
  - Edgewood, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Clinton, Maryland
  - Salisbury, Maryland
  - Silver Spring, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Lansing, Michigan
  - Marquette, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - Robbinsdale, Minnesota
  - Rochester, Minnesota
  - Saint Louis Park, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Morristown, New Jersey
  - Ocean Township, New Jersey
  - Albuquerque, New Mexico
  - Garden City, New York
  - Huntington, New York
  - Manhasset, New York
  - New York, New York
  - Poughkeepsie, New York
  - Utica, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Danville, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Kingsport, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Plano, Texas
  - The Woodlands, Texas
  - Burlington, Vermont
  - Spokane, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Belgium (2):
  - Leuven
  - Yvoir
- Canada (4):
  - Calgary
  - Kingston
  - Montreal
  - Québec
- France (5):
  - Clermont-Ferrand
  - La Rochelle
  - Montpellier
  - Nantes
  - Pringy
- Germany (7):
  - Aachen
  - Cologne
  - Essen
  - Hanover
  - Homburg
  - Tübingen
  - Ulm
- Italy (2):
  - Milan
  - Reggio Emilia
- Kuala Lumpur, Malaysia
- Netherlands (4):
  - Eindhoven
  - Maastricht
  - Nieuwegein
  - Rotterdam
- Belgrade, Serbia
- Seoul, South Korea
- Spain (2):
  - A Coruña
  - Palma de Mallorca
- Skövde, Sweden
- United Kingdom (4):
  - Birmingham
  - Liverpool
  - Manchester
  - Middlesbrough